CLINICAL TRIAL: NCT05897229
Title: Palliative Care in Patients With COVID-19: Analysis of Costs of Hospitalization in Wards and Intensive Care Units
Status: Not yet recruiting | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Ricardo Tavares de Carvalho, Collaborator Professor, Palliative Care Departament Coordinator, University of Sao Paulo General Hospital
Other Study IDs: 31385420.6.1001.0068
Record Dates: First submitted 2023-06-07; First posted 2023-06-09 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: COVID-19; Palliative Care
Keywords: Palliative care; COVID-19; Cost allocation; Cost control; Organization and Administration
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PC - end-stage disease criteria and high risk of death from the disease prior to COVID-19: Patients with severe forms of COVID-19 (RT-PCR+) admitted to a high-complexity hospital.
  Of these, patients with end-stage disease criteria and high risk of death from the disease prior to COVID-19 were admitted, at clinical criteria, to palliative care unit.
  If there are patients who received both types of treatment, this group will also be analyzed.
  Interventions: Other: Analysis of costs with patient care during hospitalization
- ICU - end-stage disease criteria and high risk of death from the disease prior to COVID-19: Patients with severe forms of COVID-19 (RT-PCR+) admitted to a high-complexity hospital.
  Of these, patients with end-stage disease criteria and high risk of death from the disease prior to COVID-19 were admitted, at clinical criteria, to the ICU.
  If there are patients who received both types of treatment, this group will also be analyzed.
  Interventions: Other: Analysis of costs with patient care during hospitalization
- PC & ICU - end-stage disease criteria and high risk of death from the disease prior to COVID-19: Patients with severe forms of COVID-19 (RT-PCR+) admitted to a high-complexity hospital.
  Of these, patients with end-stage disease criteria and high risk of death from the disease prior to COVID-19 were admitted, at clinical criteria, to the ICU and palliative care unit.
  If there are patients who received both types of treatment, this group will also be analyzed.
  Interventions: Other: Analysis of costs with patient care during hospitalization

INTERVENTIONS:
Other: Analysis of costs with patient care during hospitalization — Analysis of direct costs with supplies, medications, diets, laboratory tests and imaging exams, and invasive procedures such as mechanical ventilation, dialysis, and the use of vasoactive drugs.-analysis of costs referring to working hours of physicians, nurses and physical therapists in each unit normalized for the same number of beds.- cost minimization and consequential cost analysis.

SUMMARY:
The confrontation of COVID-19 foreshadowed a serious crisis of scarce health resources worldwide. To assist in this confrontation, the Palliative Care Scientific Technical Core of the Clinical Hospital, School of Medicine, Sao Paulo University (USP) elaborated a Triage Protocol for Palliative Care (PALI-COVID Tool) and it was possible to categorize the patients in three groups, according to the risk of death and needs of Palliative Care (PC), through the clinical evaluation of the patient that also directed them to the hospitalization resource according to their need (ward x ICU).

DETAILED DESCRIPTION:
The patients grouped as with higher risk of death and PC needs (green group) by PALI-COVID Tool were those with a profile of end-of-life, signs of clinical deterioration and risk of death on admission and thus indicated for admission to the COVID-19 Palliative Care Inpatient Unit, however some were admitted to the ICU. Objective: to analyze the direct costs of hospitalization of COVID-19 Palliative Care patients in Palliative Care Inpatient Unit and ICU screened as green group by the COVID-19 Screening Protocol developed in the institution. Methods: observational, cross-sectional and retrospective study of the service database of patients over 18 years of age screened as the green group (PALI-COVID). The variables to be investigated are related to sociodemographic and clinical data, length of stay and hospitalization scenarios, time to call for PC, outcome and costs.

ELIGIBILITY:
Inclusion Criteria:

* inpatients with severe forms of COVID-19 between April 08 and July 31, 2020
* positive reverse-transcriptase polymerase chain reaction (RT-PCR).
* patients with terminal illness and high clinical risk of death before COVID-19.
* those admitted to an ICU or palliative care unit.

Exclusion Criteria:

* absence of hospitalization cost data in the institution's electronic records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A screening protocol was created by us for stratification of patients admitted due to risk of death and PC needs - the PALICOVID. Patients classified by PALICOVID in the most severe group (terminal illness and clinical criteria of high risk of death prior to COVID-19) were referred to the PC Inpatient Unit. These patients were admitted, at the physician's discretion, in the PC unit or ICU. The mortality of patients in both groups was similar. Thus, the characterization of the sample according to demographic, clinical data, and comparative analysis of direct and indirect costs during hospitalization between the subgroups (PC, ICU and PC & ICU ) will be performed.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Direct costs (supplies) | Hospitalizations between April 8th to July 31th, 2020
  costs related to supplies, medications, diets, laboratory tests, imaging exams, and invasive procedures (such as mechanical ventilation, dialysis, and the use of vasoactive drugs). The costs will be calculate for the three groups and compared between them.
Direct costs (working hours) | Hospitalizations between April 8th to July 31th, 2020
  costs referring to working hours of health professionals (physicians, nurses and physical therapists) in each unit normalized for the same number of beds. The costs will be calculate for the three groups and compared between them.
Cost minimization, and consequential cost analysis | Hospitalizations between April 8th to July 31th, 2020
  all the costs will be compared between them to do a cost-effectiveness analysis as the death rate will be probabily similar in the three groups.

SECONDARY OUTCOMES:
Sociodemographic profile | Hospitalizations between April 8th to July 31th, 2020
  age and sex to identify and analyze the profile of the patients included in the study.
Clinical profile | Hospitalizations between April 8th to July 31th, 2020
  diagnosis, underlying disease, comorbidities to identify and analyze the profile of the patients included in the study.
Length of stay and inpatient settings | Hospitalizations between April 8th to July 31th, 2020
  length of stay at Palliative Care unit (PC), ICU and PC & ICU to identify and analyze the profile of the patients included in the study and analyze the costs.
Time to call Palliative Care group | Hospitalizations between April 8th to July 31th, 2020
  admission to the institution, date of call of PC, first assessment of PC, indication of transfer to a COVID-19 PC unit, and date of transfer to PC unit to identify and analyze the time it took for staff to recognize the need for CP for the patients that has repercussions on the cost of hospitalization.
Life-sustaining procedures | Hospitalizations between April 8th to July 31th, 2020
  such as mechanical ventilation, dialysis, and the use of vasoactive drugs to identify and analyze the use of life-sustaining procedures in the study population and analyze the costs.
Inpatient daily rates | Hospitalizations between April 8th to July 31th, 2020
  rates for Palliative Care unit (PC), ICU and PC & ICU to analyze the costs.
Outcome of hospitalization | Hospitalizations between April 8th to July 31th, 2020
  hospital discharge, transference, and death to identify and analyze the profile of the patients included in the study and to make a cost-effectiveness analysis with the all costs that will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo T de Carvalho, MD, PhD, Principal Investigator — University of Sao Paulo General Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anagusko SS, Rosa IB, Angelo MFF. Fundamentos dos Cuidados Paliativos aplicados à pandemia. In: Daniel Battacini Dei Santi, Luciana Suely Barros Cavalcante, Ednalda Maria Franck,Ricardo Tavares de Carvalho. (Org.). Cuidados Paliativos na Prática Clínica em Tempos de COVID-19. 1ed.Rio de Janeiro: Atheneu, 2021, v. 1, p. 5-15.
- [Background] Carvalho RT, Crispim DH, Franck EM, Dei Santi DB, Anagusko SS, Fukuda MV, Cavalcante LSB, Jales SMDCP, Queiroz MEG, Bonfa ESDO. Palliative care in the COVID-19 pandemic: Strategy of HCFMUSP. Clinics (Sao Paulo). 2022 Jan-Dec;77:100050. doi: 10.1016/j.clinsp.2022.100050. Epub 2022 May 17. No abstract available. PMID 35662009
- [Background] Downar J, Seccareccia D; Associated Medical Services Inc. Educational Fellows in Care at the End of Life. Palliating a pandemic: "all patients must be cared for". J Pain Symptom Manage. 2010 Feb;39(2):291-5. doi: 10.1016/j.jpainsymman.2009.11.241. PMID 20152591
- [Background] Fadul N, Elsayem AF, Bruera E. Integration of palliative care into COVID-19 pandemic planning. BMJ Support Palliat Care. 2021 Mar;11(1):40-44. doi: 10.1136/bmjspcare-2020-002364. Epub 2020 Jun 11. PMID 32527790
- [Background] Franck EM, Jales SMCP, Dei Santi DB, Cavalcante LSB, Silva MLF. A equipe multiprofissional na pandemia: novas formas de atuação, antigos desafios. In: Daniel Battacini Dei Santi, Luciana Suely Barros Cavalcante, Ednalda Maria Franck, Ricardo Tavares de Carvalho. (Org.). Cuidados Paliativos na Prática Clínica em Tempos de COVID-19. 1ed.Rio de Janeiro: Atheneu, 2021, v. 1, p. 31-44.
- [Background] May P, Normand C, Cassel JB, Del Fabbro E, Fine RL, Menz R, Morrison CA, Penrod JD, Robinson C, Morrison RS. Economics of Palliative Care for Hospitalized Adults With Serious Illness: A Meta-analysis. JAMA Intern Med. 2018 Jun 1;178(6):820-829. doi: 10.1001/jamainternmed.2018.0750. PMID 29710177
- [Background] Medical guidelines for determining prognosis in selected non-cancer diseases. The National Hospice Organization. Hosp J. 1996;11(2):47-63. doi: 10.1080/0742-969x.1996.11882820. No abstract available. PMID 8949013
- [Background] Sheridan PE, LeBrett WG, Triplett DP, Roeland EJ, Bruggeman AR, Yeung HN, Murphy JD. Cost Savings Associated With Palliative Care Among Older Adults With Advanced Cancer. Am J Hosp Palliat Care. 2021 Oct;38(10):1250-1257. doi: 10.1177/1049909120986800. Epub 2021 Jan 11. PMID 33423523
- See also: Brazil.Law No. 13.709 General Law for the Protection of Personal Data (LGPD). 2018. — http://www.planalto.gov.br/ccivil_03/_ato2015-2018/2018/lei/l13709.htm
- See also: World Health Organization(WHO).Building integrated Palliative Care programs and services.2017 — http://www.thewhpca.org/resources/category/building-integrated-palliative-care-programs-and-services
- See also: Oxford University.Our world in data: coronavirus (COVID-19) data. 2020 — http://ourworldindata.org/covid-deaths
- See also: WHO.Integrating palliative care and symptom relief into the response to humanitarian emergencies and crises: a WHO guide. 2022 — http://www.who.int/publications/i/item/9789241514460